CLINICAL TRIAL: NCT05634538
Title: Robotically Assisted PCI in Ostial Lesions
Brief Title: The ROB-OSTIAL Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor strategic decision
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104-13191
Record Dates: First submitted 2022-11-17; First posted 2022-12-02 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Ostial Lesion; Robotic-assisted PCI; PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic-assisted PCI with Corpath GRX® System (Active Comparator): Percutaneous coronary intervention (PCI) using the Corpath GRX System.
  Interventions: Device: Robotic-assisted PCI with Corpath GRX® System
- Standard PCI (Active Comparator): Percutaneous coronary intervention (PCI) using manual techniques. This arm will be completed without robotic assistance.
  Interventions: Procedure: Standard PCI

INTERVENTIONS:
Device: Robotic-assisted PCI with Corpath GRX® System — The CorPath GRX System is intended for use in the remote delivery and manipulation of guidewires and rapid exchange catheters, and remote manipulation of guide catheters during percutaneous coronary interventions (PCI).
  Arms: Robotic-assisted PCI with Corpath GRX® System
Procedure: Standard PCI — Percutaneous coronary intervention (PCI) is a procedure used to treat the blockages in a coronary artery; it opens up narrowed or blocked sections of the artery, restoring blood flow to the heart. This arm will be completed without robotic assistance.
  Arms: Standard PCI

SUMMARY:
The purpose of this study is to compare the accuracy of robotic-assisted percutaneous coronary intervention (PCI) using the CorPath GRX® System, versus standard PCI when treating ostial lesions.

CorPath GRX System (the Device) is a robotic-like device that is cleared for the remote delivery and control of heart catheterization devices. It helps doctors insert and move heart catheters (a thin, flexible tube) and similar types of devices inside patients blood vessels to treat the blockage in their heart.

The results will help to evaluate whether procedures using the CorPath GRX result in more accurate stenting (placing of a tube to keep heart vessel open) compared to standard PCI.

DETAILED DESCRIPTION:
To assess accuracy of robotic-assisted PCI in obtaining full ostial lesion coverage and minimal protrusion compared to standard PCI.

Robotically assisted PCI offers the opportunity of performing minimal device movements (up to a minimum of 1 mm) in a stable and reproducible setting. This feature may be of great help when dealing with ostial lesions, whose treatment requires a precise stent positioning to avoid strut protrusion but also geographic miss of the lesion. Robotic-assisted PCI for ostial lesions showed encouraging results in large observational registries, but no study compared this approach with standard PCI.

The aim is to perform a randomized (1:1) study comparing standard (n=33) and robotic-assisted PCI (n=33) in obtaining full lesion coverage when treating ostial lesions (ostial left main will be excluded).

Primary endpoint of the study will be full ostial coverage as assessed by IVUS imaging, while secondary endpoints will be procedural success, vessel damage and number of protruding struts in the donor vessel as assessed by IVUS imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female aged ≥18 years
* Coronary OSTIAL lesion suitable for percutaneous coronary intervention (PCI)
* The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

* Cardiogenic shock or hemodynamic instability requiring support.
* ST-elevation myocardial infarction.
* Ongoing acute renal failure.
* In the opinion of the investigator, the subject is deemed unsuitable for robotic PCI due to clinical status and/or anatomic characteristics
* More than one lesion to be treated
* Ostial left main disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Cecilia Hospital, Cotignola, RA, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic-assisted PCI With Corpath GRX® System | Standard PCI
Started | 1 (One subject was consented and randomized to the Robotic-assisted PCI arm. However, this subject was not treated with the device due severe vessel tortuosity.) | 0
Completed | 0 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject was enrolled and randomized to Robotic-assisted PCI with Corpath GRX® System, however they were withdrawn before they could be treated with the CorPath GRX due to tortuous vessel anatomy. The study was then closed and no other subjects were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic-assisted PCI With Corpath GRX® System | Standard PCI | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Count of Participants; unit: Participants] | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  Italy | 1 |  | 1
Canadian Cardiovascular Society (CCS) Angina Grade [Number; unit: units on a scale] — I:Ordinary physical activity (OPA) does not cause angina, such as walking/climbing stairs. Angina occurs with strenuous/rapid/prolonged exertion 2: Slight limitation of OPA. Angina occurs with quick/uphill walking, after meals, in cold/wind, under stress, or soon after waking. Walking >2 flat blocks & climbing >1 flight of stairs at a normal pace/conditions 3: Marked limitations of OPA. Angina occurs on walking 1-2 blocks on the level and climbing 1 flight of stairs in normal conditions/pace 4: Inability to carry on any physical activity without discomfort: angina may be present at rest
  units on a scale | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Full Ostial Coverage at Angiographic and IVUS Assessment
Description: Procedure-dependent geographic miss in millimeters (mm) obtained using intravascular ultrasound (IVUS)
Time Frame: Measured at end of procedure
Population: One subject was enrolled and randomized, but was not treated per protocol due to tortuous vessel anatomy. No IVUS information collected.
Arm/Group | Robotic-assisted PCI With Corpath GRX® System | Standard PCI
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Distance From Most Proximal Stent Strut and Coronary Ostium (mm), as Assessed by IVUS
Description: Distance from most proximal stent strut and coronary ostium (mm), as assessed by IVUS
Time Frame: Measured at end of procedure
Population: as for outcome 1
Arm/Group | Robotic-assisted PCI With Corpath GRX® System | Standard PCI
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Comparison of Participants With In-hospital Major Cardiovascular Events
Time Frame: Measured at discharge or 72 hours, whichever comes first
Population: Analysis population of the one subject enrolled and randomized.
Measure: Number; unit: Adverse Events
Arm/Group | Robotic-assisted PCI With Corpath GRX® System | Standard PCI
Number analyzed (Participants) | 1 | 0
Adverse Events | 0 |

4. Secondary Outcome: Procedural Duration
Description: Defined as the duration from when the sheath is inserted until it is removed
Time Frame: Measured at end of procedure
Population: One subject was enrolled and randomized, but was not treated per protocol due to tortuous vessel anatomy.
Measure: Number; unit: minutes
Arm/Group | Robotic-assisted PCI With Corpath GRX® System | Standard PCI
Number analyzed (Participants) | 1 | 0
minutes | 75 |

5. Secondary Outcome: Major Adverse Cardiovascular Events at 1 Month Follow-up
Time Frame: Measured at 1 month
Population: One subject was enrolled and randomized, but was not treated per protocol due to tortuous vessel anatomy. Study was shut down and no further follow-up completed.
Arm/Group | Robotic-assisted PCI With Corpath GRX® System | Standard PCI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was ascertained on the the day of the one subject enrollment. After the subject was unable to undergo the study treatment per protocol the study was discontinued due to Sponsor business decision and therefore no additional adverse event data was collected.
Description: The protocol utilized MEDDEV 2.7/3rev. 3 May 2015 ; ISO 14155:2011 for adverse event definitions.
Arm/Group | Robotic-assisted PCI With Corpath GRX® System | Standard PCI
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT05634538/Prot_SAP_000.pdf